CLINICAL TRIAL: NCT01768598
Title: An Investigation Into Risk Taking Behaviour, Bone Microstructure and Fracture Between the Sexes: What Underpins Fracture in Boys Compared to Girls During Growth?
Brief Title: Risk Taking and Fracture Study
Status: Completed | Type: Observational
Sponsor: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Heather McKay, Principal Investigator, University of British Columbia
Organization: University of British Columbia (Other)
Other Study IDs: H10-00044
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Fracture
Keywords: Wrist Fracture; Adolescents; Risk Taking Behaviour; Bone Microstructure
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Fracture - Boys: Boys who have sustained a distal radius fracture
  Interventions: Other: Fracture - Boys
- Fracture - Girls: Girls who have sustained a distal radius fracture
  Interventions: Other: Fracture - Girls
- Non Fracture - Boys: Boys who have not sustained a distal radius fracture
  Interventions: Other: Non Fracture - Boys
- Non Fracture - Girls: Girls who have not sustained a distal radius fracture
  Interventions: Other: Non Fracture - Girls

INTERVENTIONS:
Other: Fracture - Boys — Annual measurements of risk taking behaviour, body composition, bone microstructure, balance, diet, and physical activity over 4 years
  Groups: Fracture - Boys
Other: Fracture - Girls — Annual measurements of risk taking behaviour, body composition, bone microstructure, balance, diet, and physical activity over 4 years
  Groups: Fracture - Girls
Other: Non Fracture - Boys — Annual measurements of risk taking behaviour, body composition, bone microstructure, balance, diet, and physical activity over 4 years
  Groups: Non Fracture - Boys
Other: Non Fracture - Girls — Annual measurements of risk taking behaviour, body composition, bone microstructure, balance, diet, and physical activity over 4 years
  Groups: Non Fracture - Girls

SUMMARY:
Boys suffer a disproportionately large number of fractures compared to girls (55-60%). This study aims to determine why this is the case by identifying risk factors for wrist fractures. The increase in fracture during childhood and adolescence may be associated with 1) risk-taking behaviour in boys, 2) obesity trends in boys during childhood and adolescence, and/or 3) impaired acquisition of bone strength during childhood and adolescence. Importantly from a knowledge translation perspective, modifiable factors such as behaviour, dietary habits or physical activity in boys may predict fracture.

The investigators will measure 400 children (100 girls and 100 boys who have sustained a fracture; 100 same age and sex friends) across 4 years of growth. This study will assess risk behaviours, diet, physical activity, motor proficiency (i.e., balance and coordination), fat and muscle mass and bone strength to determine if there are, 1) differences in whether all or some of these factors predict fractures in boys compared with girls and, 2) whether these factors track forward similarly in boys compared with girls as children advance through the growth spurt.

DETAILED DESCRIPTION:
The investigators aim to better characterize factors that contribute to fracture in boys and girls and to assess whether such factors track across a four year period. The innovation is to use novel methods and an integrated approach, to measure the influence of risk-taking behaviour, body composition, bone microstructure, motor proficiency, diet and physical activity in one model across growth. This will provide a more comprehensive picture of the key multi-factorial predictors of fracture within- and between-sexes. This essential information will provide the basis for change in public health policy, clinical practice, community programs, and targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* Boys aged 9-15 and Girls aged 8-13
* Fracture to distal radius after low to moderate energy trauma
* No other health concerns
* Healthy (non fracture) subjects for comparison

Exclusion Criteria:

* Fracture is a result of severe trauma
* Children with ontological medical conditions

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fracture patients will be recruited from the orthopaedic clinic at BC Children's Hospital.
  Non-fracture subjects will be recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Characterization of factors that contribute to fractures in boys and girls | Baseline (<3 months after injury)
  The factors include:
  1. Risk taking behaviour - protection motivation variables, anticipated regret and excitement and impulsivity dispositions
  2. Body composition - total body mass, fat mass, lean mass
  3. Bone microstructure - cortical and trabecular bone outcomes
  4. Dietary intake - calcium
  5. Physical activity

SECONDARY OUTCOMES:
Tracking of Risk Factors | 4 years
  The outcomes will be measured across a 3 year interval (4 years in total) to determine whether factors track similarly in boys compared with girls over time and to assess their continued (or not) contribution to fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Heather McKay, PhD, Principal Investigator — Centre for Hip Health and Mobility
Locations (2):
- Canada (2):
  - Centre for Hip Health and Mobility, Vancouver, British Columbia
  - British Columbia Children's Hospital, Vancouver, British Columbia